CLINICAL TRIAL: NCT03838380
Title: Peripartum Management of Gestational Diabetes Using a Digital Healthcare Service: a Pilot, Randomized Controlled Study
Brief Title: Smartphone Application for the Management of Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Cheol-Young Park, Professor, Division of Endocrionology and metabolism, Department of Internal medicine, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KBSMC2016-11-049
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional management group (No Intervention): The conventional management group received standard GDM management and could freely use the smartphone healthcare application.
- mobile management group (Experimental): The mobile management group received mobile healthcare services through smartphone application specifically developed for this trial including tailored mobile coaching.
  Interventions: Other: Smartphone application

INTERVENTIONS:
Other: Smartphone application — Mobile management group participants were given monitoring system devices including a glucometer with Bluetooth connectivity and an accelerometer to detect physical activity level. The mobile phone application specifically designed for this study was installed at enrollment for the mobile management group to collect clinical data and messages from the patients. The application consisted of four sections: clinical data, nutrition and diet, medication, and messaging system and information. Patients allocated to the mobile management group recorded their blood glucose level and diet via the smartphone application, and health care providers regularly scanned clinical data and messages from patients and sent return messages with tailored medical and nutritional guidance.
  Arms: mobile management group

SUMMARY:
The prevalence of gestational diabetes mellitus (GDM) has been progressively increasing. It is important to recognize and treat GDM to minimize the risk of maternal and neonatal complications. Multifaceted professional interventions are effective in the management of GDM and mobile healthcare can be an effective approach. The purpose of the current study was to develop and evaluate a model for prevention and management of GDM using mobile healthcare. Subjects with no previous history of diabetes, who were diagnosed with GDM during 24-28 weeks of gestation, were randomly divided into a conventional management group and a mobile management group. The conventional mangement group received conventional GDM management and could freely use the mobile healthcare application. The mobile management group received mobile healthcare services including tailored mobile coaching. The effectiveness of the management using the application were evaluated through the result values of the laboratory tests, anthropometric measurement performed during the study period and perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnant women diagnosed as GDM at 24 to 28 weeks of gestation were included.

Exclusion Criteria:

* Patients after 30th week of gestation and patients with pregestational diabetes were excluded from participating in the study. Patients who were unable to understand Korean, were unfamiliar with mobile phones, who did not have access to a mobile phone, or who were already receiving services from another mobile healthcare agency were also excluded.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
hemoglobin A1c levels | up to 4 to 12weeks after delivery
  serum glycated hemoglobin levels

SECONDARY OUTCOMES:
body weight | up to 4 to 12weeks after delivery
  the changes in body weight
body mass index | up to 4 to 12weeks after delivery
  the changes in body mass index
percent body fat | up to 4 to 12weeks after delivery
  the changes in percent body fat
HOMA IR(homeostatic model assessment insulin resistance) | up to 4 to 12weeks after delivery
  the changes in insulin resistance
HOMA-ß (homeostatic model assessment ß-cell dysfunction ) | up to 4 to 12weeks after delivery
  the changes in ß-cell dysfunction
Neonate large for gestational age | at the day of delivery
  Birth weight of neonates of GDM patients
Mode of delivery | at the day of delivery
  Rate of cesarean section

CONTACTS AND LOCATIONS:
Locations (1):
- Kangbuk Samsung hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sung JH, Lee DY, Min KP, Park CY. Peripartum Management of Gestational Diabetes Using a Digital Health Care Service: A Pilot, Randomized Controlled Study. Clin Ther. 2019 Nov;41(11):2426-2434. doi: 10.1016/j.clinthera.2019.09.005. Epub 2019 Oct 4. PMID 31587813